CLINICAL TRIAL: NCT02497703
Title: Interactive Exoskeleton Robot for Walking - Knee Joint
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Chinese University of Hong Kong (Other)
Collaborators: The Hong Kong Polytechnic University (Other)
Responsible Party: Principal Investigator, Raymond KY Tong, Professor, Chinese University of Hong Kong
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2015.037T (Knee)
Record Dates: First submitted 2015-07-12; First posted 2015-07-14 (Estimated); Last update posted 2017-09-18 (Actual); Status verified 2017-09

CONDITIONS: Stroke
MeSH Terms: conditions — Stroke

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Knee robot (Experimental): This robotic system has been developed to facilitate functional motor recovery by practices walking with a one joint motor powered exoskeleton
  Interventions: Device: Knee robot

INTERVENTIONS:
Device: Knee robot

SUMMARY:
An exoskeleton robotic knee system for stroke rehabilitation is proposed in this study. This robotic system has been developed to facilitate functional motor recovery by practices walking with a one joint motor powered exoskeleton to reduce the muscle weakness in the shank and reduce the hyperextension in the knee joint. The robotic knee system is able to sense the gait pattern from the stroke patients and assist the walking and control the knee angle. The clinical trial will use repeated measurements to evaluate the effectiveness of the robotic knee system in gait rehabilitation post stroke.

ELIGIBILITY:
Inclusion Criteria:

1. Ischemic or hemorrphagic stroke with drop foot problem.
2. Sufficient cognition to follow simple instructions and to understand the content and purpose of the study. (Mini-Mental State Examination > 20)
3. Capable of standing and walking independently for an extended period of time. (Functional Ambulation Category > 3, Berg Balance Scale > 40)

Exclusion Criteria:

1. Any medical or psychological dysfunctions that would affect their ability to comply with test study protocol, such as lower back pain, neuralgia, rotational vertigo, muscloskeletal disorders, injuries, and pregnancy.
2. Any severe contractures in hip, knee, or ankle joint that would preclude passive range of motion in the lower extremity.
3. Participation in any therapeutic treatment ("outside therapy") performed with the lower extremity during the planned study, including the baseline and the followup.

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Actual)
Dates: Start 2015-05-27 (Actual); Primary Completion 2016-10-14 (Actual); Study Completion 2016-12-31 (Actual)

PRIMARY OUTCOMES:
Functional Ambulation Category | 3-month followup
  Patients can be rated on the following categories:
  0: Patient cannot walk, or needs help from 2 or more persons
  1. Patients needs firm continuous support from 1 person who helps carrying weight and with balance
  2. Patient needs continuous or intermittent support of one person to help with balance and coordination.
  3. Patient requires verbal supervision or stand-by help from one person without physical contact
  4. Patient can walk independently on level ground, but requires help on stairs, slopes or uneven surfaces
  5. Patient can walk independently anywhere
6-minute Walk Test | 3-month followup
  Walk as far a distance as possible over 6 minutes with their preferred speed; assistive devices can be used but kept consistent from test to test Individual should be able to ambulate without physical assistance.

SECONDARY OUTCOMES:
Kinematic and Kinetic Gait Motion Capture | 3-month followup
  Motion analysis to evaluation the ankle, knee and hip angles; and ground reaction force
Fugl-Meyer Assessment Lower Extremity | 3-month followup
  Evaluates and measures motor function recovery in post-stroke hemiplegic patients Used in both clinical and research settings, maximum score = 34
Timed 10-meter Walk Test | 3-month followup
  The individual is instructed to walk a set distance (10 meters). Time is measured while the individual walks the set distance (often the individual is given space to accelerate to his/her preferred walking speed (this distance is not included when determining speed). The distance covered is divided by the time it took the individual to walk that distance.
Modified Ashworth Scale | 3-month followup
  Tests resistance to passive movement about a joint with varying degrees of velocity; scores range from 0-4, with 6 choices
Berg Balance Scale | 3-month followup
  Static and dynamic activities of varying difficulty are performed Item-level scores range from 0-4, determined by ability to perform the assessed activity Item scores are summed Maximum score = 56

CONTACTS AND LOCATIONS:
Locations (2):
- Hong Kong (2):
  - Department of Biomedical Engineering, The Chinese University of Hong Kong, Hong Kong
  - Interdisciplinary Division of Biomedical Engineering. The Hong Kong Polytechnic Univesity, Hong Kong